CLINICAL TRIAL: NCT00922285
Title: Art Therapy Interventions With Caregivers Supporting Pediatric Patients Who Are Undergoing Bone Marrow Transplantation for Cancer
Brief Title: Art Therapy for Caregivers of Young Patients Undergoing Bone Marrow Transplant for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 08028; P30CA033572 (NIH); CHNMC-08028; CDR0000642781 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Health Status Unknown; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; health status unknown
MeSH Terms: interventions — Psychiatric Rehabilitation; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Art Therapy (Experimental)
  Interventions: Other: psychosocial support for caregiver; Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: stress management therapy

INTERVENTIONS:
Other: psychosocial support for caregiver — 6 weekly 60 minute sessions
Other: questionnaire administration — Evaluated at baseline, week 1 and week 6 of art therapy
Procedure: quality-of-life assessment — Evaluated at baseline, week 1 and week 6 of art therapy
Procedure: stress management therapy — 6 weekly 60 minute sessions

SUMMARY:
RATIONALE: Art therapy may help relieve emotional distress in caregivers of young patients undergoing bone marrow transplant for cancer.

PURPOSE: This clinical trial is studying art therapy for caregivers of young patients undergoing bone marrow transplant for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Test the effects of an art therapy intervention on emotional distress in caregivers of pediatric patients undergoing bone marrow transplantation for cancer.
* Describe pro-social interactions of caregivers of pediatric patients undergoing bone marrow transplantation for cancer.
* Describe the illness experience of caregivers and how it is impacted by the art therapy intervention.
* Describe the caregivers' current health-related quality of life and life meaning prior to pediatric patients initiation of bone marrow transplantation for cancer.
* Determine the effect size for calculating the sample needed for a randomized clinical trial.

OUTLINE: Caregivers undergo art therapy over 60 minutes once a week for 6 weeks. Each session comprises developing trust through the expression of support, affirmation, and collaboration; creating intimacy through attunement; exploring affective states; integrative processing through the creation of an autobiographical narrative; and identifying opportunities for continued exploration and resources that support the client, should that exploration become necessary.

Caregivers also complete a Meaning of Life Questionnaire and a Family Quality of Life Scale at baseline and at the end of week 6.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Family caregiver identified by the patient's physician as most involved in the patient care including, but not limited to, the following:

  * Mother
  * Father
  * Grandmother
  * Grandfather
  * Aunt
  * Uncle
  * Older sibling
* One caregiver per pediatric patient
* No caregivers who are part of an institutional system and are temporarily fulfilling the custodial role of the patient (i.e., foster parents)

PATIENT CHARACTERISTICS:

* Able to speak and read English and/or Spanish
* No uncontrolled mental health and/or physical condition

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Emotional distress | Baseline, week 1 and week 6 of art therapy
Pro-social interactions | Baseline, week 1 and week 6 of art therapy
Illness experience of caregivers and how it is impacted by the art therapy intervention | Baseline, week 1 and week 6 of art therapy
Caregivers' current health-related quality of life and life meaning | Baseline, week 1 and week 6 of art therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kate Kravits, RN, MA, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States